CLINICAL TRIAL: NCT05269108
Title: Safety and Efficacy of Fluoroscopy-free Technique During Retrograde Intrarenal Surgery for Renal Stones: A Prospective, Randomized, Non-inferiority Trial
Brief Title: Safety and Efficacy of Fluoroscopy-free Technique During Retrograde Intrarenal Surgery for Renal Stones
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Abul-fotouh Ahmed, Professor, Al-Azhar University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Uro_Azhar_2_022
Record Dates: First submitted 2022-02-25; First posted 2022-03-07 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Kidney Calculi; Radiation Exposure; Retrograde Intrarenal Surgery
MeSH Terms: conditions — Kidney Calculi

STUDY DESIGN:
Intervention Model Description: The 1st group: Fluoroscopy-free RIRS. The 2nd group: Fluoroscopy-guided RIRS.
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fluoroscopy-free RIRS (Experimental): Patients will be treated by RIRS without fluoroscopy
  Interventions: Procedure: Fluoroscopy-free RIRS
- Standard RIRS (Active Comparator): Standard RIRS under fluoroscopy-guidance will be performed
  Interventions: Procedure: Standard RIRS

INTERVENTIONS:
Procedure: Fluoroscopy-free RIRS — RIRS for renal stone under direct visualization, without fluoroscopy
  Arms: Fluoroscopy-free RIRS
Procedure: Standard RIRS — RIRS for renal stone under fluoroscopy-guidance
  Arms: Standard RIRS

SUMMARY:
Aiming to reduce radiation exposure to patients and physicians, the investigators conduct this study protocol to evaluate the possibility of performing retrograde intrarenal surgery (RIRS) under direct visualization without fluoroscopy. the investigators will prospectively evaluate the outcome of fluoroscopy-free RIRS for renal stones in comparison with the standard technique. The investigators expected that the fluoroscopy-free technique has high safety and efficacy even in complicated cases.

DETAILED DESCRIPTION:
With improved flexible URS instrumentation and lithotripsy technology, retrograde intrarenal surgery (RIRS) became an alternative and excellent option for renal stones. Fluoroscopy imaging may be necessary during various steps of RIRS, such as insertion of a guidewire and stent, access sheath insertion, detection of stone location and size, and assessment of collecting system anatomy.

In an effort to decrease radiation exposure, several studies were conducted to evaluate the possibility of performing RIRS under direct visualization without fluoroscopy. Most studies concluded that fluoroscopy-free RIRS is a feasible, effective, and safe technique. The reported stone-free rate ranged from 83.8% to 95.7%. No major complications were observed.

Despite the reported high safety and efficacy of the fluoroscopy-free RIRS technique, most of the studies were retrospective and included only uncomplicated cases, and none of the studies address its results against control.

In the present study, the investigators will prospectively evaluate the efficacy and safety of fluoroscopy-free RIRS for renal stones in comparison with fluoroscopy-guided technique as standard control. The study will include all patients with renal stones amenable to RIRS. The investigators expected that the fluoroscopy-free technique can deal with large stones and complex situations with high safety and success rate. The study hypothesis is that "the fluoroscopy-free technique has efficacy and safety similar to the fluoroscopy-guided technique".

The investigators also aim to determine the patients and surgical characteristics impacting the need for fluoroscopy. The intra-operative fluoroscopy imaging is expected to be necessary during RIRS, especially in complicated cases. In the fluoroscopic-free group, the fluoroscopic equipment will be available in the operating room and will be used if needed.

ELIGIBILITY:
Inclusion Criteria:

* Renal stone.
* Stone size: ≥10 mm.

Exclusion Criteria:

* Partial and complete staghorn stones.
* Pregnant women.
* Morbid obesity.
* Uncorrectable coagulation disorders.
* Active urinary tract infection (UTI).
* Stone in a calyceal diverticulum.
* Urinary tract obstruction distal to the stone.
* Concomitant pathology that needs intervention in the same setting.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 520 (Estimated)
Dates: Start 2022-02-25 (Actual); Primary Completion 2024-02 (Estimated); Study Completion 2024-04 (Estimated)

PRIMARY OUTCOMES:
stone-free rate | 3-months after the intervention.
  defined as no residual stone or residual fragment(s) less than 4 mm (as confirmed by CT-UT).
complication rate | intraoperative till 3-months postoperative complications
  intraoperative and postoperative complications

SECONDARY OUTCOMES:
fluoroscopy time | intraoperative
  intraoperative fluoroscopy imaging
Operative time | The procedure time
  Time from induction of anesthesia till the end of the procedure
the need for fluoroscopy | Intraoperative
  The need for fluoroscopy imaging in a fluoroscopy-free group

CONTACTS AND LOCATIONS:
Overall Officials: Abul-fotouh Ahmed, MD, Principal Investigator — Al-Azhar University Hospitals, Cairo, Egypt
Locations (1):
- Urology Department, Al-Azhar University Hospital, Cairo, Egypt